CLINICAL TRIAL: NCT05669248
Title: A Follow-up Study of Immune Dysregulation in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: Qilu-20221224-pang
Record Dates: First submitted 2022-12-29; First posted 2022-12-30 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-12

CONDITIONS: COVID-19; Immunosuppression
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mid covid-19 patients: Participant is diagnosed with symptomatic COVID-19 by a positive PCR for SARS-CoV-2 or antigen quicktest and meet the standard of mild COVID-19
  Interventions: Diagnostic Test: mid covid-19 patients

INTERVENTIONS:
Diagnostic Test: mid covid-19 patients — Collect the patient's whole blood for testing

SUMMARY:
In order to detect the immunosuppression status of COVID-19 patients, this study collected blood samples of COVID-19 patients on the 10th, 20th and 30th days after the onset of symptoms, and detected the proinflammatory, anti-inflammatory factors，immunosuppressive marker，immune cells in the blood samples to evaluate the immunosuppression status of COVID-19 patients.

DETAILED DESCRIPTION:
After SARS-CoV-2 infection, the patient's immune system is overactivated. While the immune cells release a large number of proinflammatory factors, anti-inflammatory response starts at the same time. Anti-inflammatory factors such as IL-4, IL-10, and IL-37 will be compensated to resist the release of proinflammatory factors and prevent the further development of systemic inflammatory response. However, when the anti-inflammatory factor is excessively released, it will cause compensatory response syndrome, leading to immunosuppression. Whether the level of anti-inflammatory factors continues to rise, and whether it will lead to the persistence of later immunosuppression is unknown. Therefore, this study intends to recruit COVID-19 patients, detect the pro-inflammatory and anti-inflammatory factors，immunosuppressive marker，immune cells in 10 days, 20days, and 30days after the symptoms appear, and evaluate the immunosuppression status of patients with COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Participant is diagnosed with symptomatic COVID-19 by a positive PCR for SARS-CoV-2 or antigen quicktest.
2. Study participant is 18 years of age or older

Exclusion Criteria:

1. Patients with immunosuppression, including HIV infection, hematopoietic stem cell transplantation and high-dose immunosuppressant therapy
2. Pregnancy or breastfeeding
3. Patients receiving chemotherapy or other cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant is diagnosed with symptomatic COVID-19 by a positive PCR for SARS-CoV-2 or antigen quicktest.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The concentration of inflammatory markers (IL-1β、IL-2、 IL-2R 、IL-4 、 IL-6 、 IL-8、 IL-10 、IFN-γ、TNF-α 、VEGF, etc.) in peripheral blood. | 10, 20, 30days
The concentration of immunosuppression makers(HLA-DR, PD-1, TIM-3,etc.) in peripheral blood. | 10, 20, 30days
The number of immune cells(Th1/Th2 cell, Treg cell, MDSCs,etc.) in peripheral blood. | 10, 20, 30days

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No